CLINICAL TRIAL: NCT03684655
Title: Imaging Immune Activation in HIV Infection
Brief Title: Imaging Immune Activation in HIV by PET-MR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CellSight Technologies, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-20302
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: HIV Infections
Keywords: HIV infection; Positron Emission Tomography; F-AraG; Magnetic Resonance Imaging
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Adults with HIV Infection taking or not taking antiretroviral therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]F-AraG (Experimental): radiofluorinated imaging agent, [18F]F-AraG (2'-deoxy-2'-fluoro-9-β-D-arabinofuranosylguanine)
  Trade name: VisAcT
  Interventions: Drug: [18F]F-AraG (2'-deoxy-2'-fluoro-9-β-D-arabinofuranosylguanine)

INTERVENTIONS:
Drug: [18F]F-AraG (2'-deoxy-2'-fluoro-9-β-D-arabinofuranosylguanine) — [18F]F-AraG is a radiolabeled high affinity substrate for deoxyguanosine kinase (dGK) and a low affinity substrate for deoxycytidine kinase (dCK), which are over-expressed in activated T cells.
  Other Names: VisAcT

SUMMARY:
This is a single center exploratory imaging study involving one intravenous microdose of [18F]F-AraG followed by whole-body positron emission tomography-magnetic resonance (PET-MR) imaging in HIV infected individuals to determine the anatomical distribution of the PET tracer. Participants will be enrolled if they were treated during early or late HIV infection. In addition, individuals not on antiretroviral therapy (ART) or with HIV-1 plasma RNA levels >5,000 copies/mL will be enrolled. Up to 30 participants will be enrolled with HIV.

DETAILED DESCRIPTION:
The PET radiofluorinated imaging agent, [18F]F-AraG (2'-deoxy-2'-fluoro-9-β-D-arabinofuranosylguanine; trade name VisAcT) localizes to sites of immune activation and is predominantly accumulated in proliferative T cells. As a result, there is interest in imaging residual immune activation in the setting of both treated and untreated HIV-1 infection, a disease in which chronic immune activation and inflammation may lead to significant morbidity, despite the use of otherwise suppressive ART.

The primary endpoint is to determine the anatomical distribution of [18F]F-AraG in HIV-infected individuals taking or not taking antiretroviral therapy.

Secondary objectives are to determine if [18F]F-AraG PET-MRI is able to detect differences in T cell activation between patients with early versus late treated HIV infection and to determine if [18F]F-AraG uptake correlates with direct blood and tissue measures of HIV reservoir size and activity in the above cohorts/studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Ability to read and understand written informed consent document
3. HIV infection, and Initiated a combination ART regimen, or, has never received ART, or, has received ART in the past, but has not been taking for a least 1 week prior to study imaging.

   (Of note, per Department of Health and Human Services (DHHS) guidelines, the protocol team will strongly recommend that all HIV+ participants initiate ART who not done so already, both for their own health and to prevent the transmission of HIV infection.)
4. Laboratory evaluations obtained within 60 days prior to entry. i. Platelet count ≥100,000/mm3 ii. ANC >1500/mm3 iii. Aspartate aminotransferase (AST) <2 x ULN iv. Alanine aminotransferase (ALT) <2 x ULN v. CD4+ T cell count >100 cells/mm3 for HIV infected individuals vi. Calculated creatinine clearance (CrCl) ≥60 mL/min as estimated by the Cockcroft-Gault equation: For men, (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dL x 72) = CrCl (mL/min)*

   * For women, multiply the result by 0.85 = CrCl (mL/min)

Exclusion Criteria:

1. Exclusion criteria will include any contra-indication to MRI, including permanent pacemaker, implantable metallic device/ prosthetic, aneurysm clip, non-removable piercing, or severe claustrophobia
2. Any medical condition that would compromise the imaging acquisition, in the opinion of the investigator
3. Individuals who have received systemic immune modifying therapy within 60 days of study enrollment (excluding HIV DNA vaccine).
4. Participants who are pregnant (female participants of childbearing age will be tested prior to injection of imaging agent at entry visit/initial visit - positive test will exclude from further participation in the study)
5. Participants who are breastfeeding
6. Female participants of reproductive potential (defined as women who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months), or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy) must have a negative urine or serum pregnancy test with a sensitivity of at least 25 mIU/mL performed at the entry/initial visit, and again within 24 hours prior to PET imaging. Females of reproductive potential will need to be on 2 forms of birth control (excluding withdrawal or timing methods).
7. Participants who have had prior allogeneic stem cell or solid organ transplant
8. Screening absolute neutrophil count <1,500 cells/mm3, platelet count <100,000 cells/mm3, hemoglobin < 8 mg/dL, estimated creatinine clearance <60 mL/minute, aspartate aminotransferase >2 x ULN, alanine aminotransferase >2 x ULN.
9. Serious illness requiring hospitalization or parental antibiotics within the preceding 3 months
10. Current HIV-related opportunistic infection such as pneumocystis pneumonia, disseminated microbacterial infection, invasive cryptococcal disease, candidal esophagitis (limited oral thrush acceptable) and cerebral toxoplasmosis
11. Previously diagnosed myelodysplasia syndrome. or history of lymphoproliferative disease prior to study entry
12. History of congestive heart failure as defined by physician documentation in the medical record at any time prior to screening that required medication for heart failure or that required medical management within 1 year prior to study entry
13. Active Hepatitis C virus (HCV) infection. Prior history of treated HCV infection with sustained virological response will be allowed.
14. Active systemic autoimmune diseases.
15. Routine clinical vaccination within 14 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Anatomical distribution of [18F]F-AraG | 1-4 hours
  Anatomical distribution of [18F]F-AraG in HIV-infected individuals taking or not taking antiretroviral therapy as determined by PET-MR imaging.

SECONDARY OUTCOMES:
[18F]F-AraG uptake in early and later-treated HIV infection | 1-4 hours
  Determine if [18F]F-AraG PET-MRI is able to detect differences in T cell activation in early versus late treated HIV infection, and between HIV infected and historical HIV-uninfected controls
Correlate [18F]F-AraG uptake with measures of HIV persistence | 1-2 weeks
  Determine if [18F]F-AraG uptake correlates with direct blood and tissue measures of HIV reservoir size and activity in the above cohorts/studies.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Henrich, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from primary and secondary outcome measures will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available 6 months following study completion.
Access Criteria: Data access requests will be reviewed by the principal investigator and study co-investigators. Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Franc BL, Goth S, MacKenzie J, Li X, Blecha J, Lam T, Jivan S, Hawkins RA, VanBrocklin H. In Vivo PET Imaging of the Activated Immune Environment in a Small Animal Model of Inflammatory Arthritis. Mol Imaging. 2017 Jan 1;16:1536012117712638. doi: 10.1177/1536012117712638. PMID 28625080
- [Background] Ronald JA, Kim BS, Gowrishankar G, Namavari M, Alam IS, D'Souza A, Nishikii H, Chuang HY, Ilovich O, Lin CF, Reeves R, Shuhendler A, Hoehne A, Chan CT, Baker J, Yaghoubi SS, VanBrocklin HF, Hawkins R, Franc BL, Jivan S, Slater JB, Verdin EF, Gao KT, Benjamin J, Negrin R, Gambhir SS. A PET Imaging Strategy to Visualize Activated T Cells in Acute Graft-versus-Host Disease Elicited by Allogenic Hematopoietic Cell Transplant. Cancer Res. 2017 Jun 1;77(11):2893-2902. doi: 10.1158/0008-5472.CAN-16-2953. PMID 28572504